CLINICAL TRIAL: NCT07207278
Title: Multi Omics Molecular Characteristics and Immunophenotyping of Lung Signet Ring Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Zhejiang University (Other); General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025ZN214-1
Record Dates: First submitted 2025-09-19; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Signet Ring Cell Carcinoma of the Lung
Keywords: LSRCC; Multi-omics analysis; Immune subtyping
MeSH Terms: interventions — alectinib; Crizotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This study was a retrospective sample analysis without patient intervention; all operations were based on archived FFPE tissues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Chinese LSRCC Multi-omics Cohort: This cohort comprises 39 treatment-naïve patients with histopathologically confirmed lung signet ring cell carcinoma (LSRCC) enrolled across multiple medical centers in China. Key molecular features include frequent mutations in core genes, distinct copy number variations (CNVs), and transcriptional up- and down-regulation of novel biomarkers. Tumor immune microenvironment (TIME) profiling classified patients into three subtypes: I, II, and III.
  Interventions: Drug: Patients with specific TIME subtype and ALK fusion mutations (confirmed via RNA-seq and OncoKB annotation) will receive tyrosine kinase inhibitors (TKIs, e.g., alectinib or crizotinib) as first-line

INTERVENTIONS:
Drug: Patients with specific TIME subtype and ALK fusion mutations (confirmed via RNA-seq and OncoKB annotation) will receive tyrosine kinase inhibitors (TKIs, e.g., alectinib or crizotinib) as first-line — Patients with specific TIME subtype and ALK fusion mutations (confirmed via RNA-seq and OncoKB annotation) will receive tyrosine kinase inhibitors (TKIs, e.g., alectinib or crizotinib) as first-line therapy. Clinical response will be assessed via RECIST v1.1 criteria using serial CT imaging (baseline, 8 weeks, and every 12 weeks thereafter). Correlative analyses will evaluate TKI efficacy in relation to TIME subtype, ALK fusion variant, and multi-omic signatures.

SUMMARY:
This study aims to reveal the molecular characteristics and immune microenvironmental profile of signet ring cell carcinoma of the lung (LSRCC) in the Chinese population through integrated multi-omics analyses. The project plans to enroll formalin-fixed paraffin-embedded (FFPE) tissue samples and paired adjacent tissues from 39 patients with previously untreated LSRCC to establish a Chinese LSRCC molecular database. Whole-exome sequencing (WES) will be used to analyze gene mutations, such as single nucleotide variants (SNVs), copy number variants (CNVs), and fusion events. RNA-seq will be used to screen for differentially expressed genes (DEGs) and perform immunophenotyping, while multiplex immunohistochemistry will be employed to quantify the tumor immune microenvironment (TIME). The successful implementation of this project is expected to identify novel molecular biomarkers specific to the Chinese LSRCC population, enhance understanding of the unique immune phenotypes within this group, and-combined with clinical follow-up-establish correlations between molecular/immune signatures and therapeutic efficacy assessments, thereby providing evidence-based medical support for subsequent personalized precision diagnosis and treatment of LSRCC in this population.

DETAILED DESCRIPTION:
This study aims to reveal the molecular characteristics and immune microenvironmental profile of signet ring cell carcinoma of the lung (LSRCC) in the Chinese population through integrated multi-omics analyses. The project plans to enroll formalin-fixed paraffin-embedded (FFPE) tissue samples and paired adjacent tissues from 39 patients with previously untreated LSRCC to establish a Chinese LSRCC molecular database. Whole-exome sequencing (WES) will be used to analyze gene mutations, including single nucleotide variants (SNVs), copy number variants (CNVs), and fusion events. RNA-seq will be utilized to screen for differentially expressed genes (DEGs) and conduct immunophenotyping, while multiplex immunohistochemistry will be applied to quantify the tumor immune microenvironment (TIME). The successful implementation of this project is expected to identify novel molecular biomarkers specific to the Chinese LSRCC population, enhance understanding of the unique immune phenotypes within this group, and-combined with clinical follow-up-establish correlations between molecular/immune signatures and therapeutic efficacy assessments, thereby providing evidence-based medical support for subsequent personalized precision diagnosis and treatment of LSRCC in this population.

ELIGIBILITY:
Inclusion Criteria:

1.Histologically confirmed, previously untreated LSRCC; 2. Adequate FFPE tumor tissue and paired adjacent non-tumor tissue available; 3. Expected survival ≥ 12 weeks; 4. Patients (or their legal guardians) willing and able to provide written informed consent; 5.Availability of complete pathology and imaging data.

Exclusion Criteria:

1. Prior systemic anticancer therapy; 2. Secondary LSRCC (i.e., metastatic signet ring cell carcinoma originating from a non-lung primary site); 3. Concurrent other malignancies; 4. Incomplete pathology results, missing imaging data, or unreliable follow-up information; 5. Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adults (≥18 years) with newly diagnosed, histopathologically confirmed lung signet ring cell carcinoma (LSRCC) who have not received prior systemic anticancer therapy. All cases must have formalin-fixed paraffin-embedded (FFPE) tissue samples available. Additional inclusion criteria include measurable disease per RECIST v1.1 on contrast-enhanced CT, ECOG performance status 0-2, and adequate organ function. Patients with concurrent malignancies, prior exposure to any ALK-targeted agent, or known contraindications to TKI therapy are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Week 8 Objective Response Rate (ORR) by RECIST v1.1 in ALK Fusion-Positive LSRCC Patients with Hybrid TIME Subtype | 8 weeks
  Objective Response Rate (ORR), defined as the proportion of patients achieving Complete Response (CR) or Partial Response (PR) per RECIST v1.1 criteria, assessed via contrast-enhanced CT at Week 8 following initiation of TKI therapy.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From baseline until disease progression or death (assessed up to 24 months).
  Time from initiation of TKI therapy to the first documented radiologic disease progression (as per RECIST v1.1) or death from any cause, whichever occurs first.
Overall Survival (OS) | From baseline until death from any cause (assessed up to 36 months).
  Time from initiation of TKI therapy to death from any cause.
Duration of Response (DoR) | From first response until progression or death (assessed up to 24 months).
  Among patients who achieve an objective response (CR or PR), the time from the first documented response to disease progression or death from any cause.
Disease Control Rate (DCR) at Week 8 | 8 weeks
  Proportion of patients achieving Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST v1.1 at Week 8.
Safety and Tolerability of TKI Therapy | From initiation of TKI therapy until 30 days after the last dose (assessed up to 24 months).
  Incidence and severity of adverse events, laboratory abnormalities, and dose modifications, graded according to NCI-CTCAE version 5.0.
Concordance Between Baseline mIHC-Defined TIME Subtypes and Treatment Outcomes | From baseline until disease progression or death (assessed up to 24 months).
  Agreement between baseline multiplex immunohistochemistry (mIHC)-defined TIME subtypes (I, II, III) and real-world treatment outcomes (ORR and PFS) across the full cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Translational Medicine, Affiliated Hangzhou First People's Hospital, Westlake University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No